CLINICAL TRIAL: NCT03480100
Title: Non-interventional Study to Investigate the Efficacy and Tolerability of Ectoin Nasal Douche (END01) in Patients With Acute Viral Rhinosinusitis
Brief Title: Non-interventional Study of Ectoin Nasal Douche (END01) in Patients With Acute Viral Rhinosinusitis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PPL-106
Record Dates: First submitted 2017-11-30; First posted 2018-03-29 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Acute Rhinosinusitis
Keywords: rhinosinusitis; nasal irrigation; nasal douche; Ectoin
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Xylometazoline Nasal spray: 1 spray per nostril as often as required but not exceeding 3 sprays per nostril per day
  Interventions: Drug: Xylometazoline Nasal Spray
- Xylometazoline + Ectoin Nasal Douche: Xylometazoline: 1 spray per nostril as often as required but not exceeding 3 sprays per nostril per day, Ectoin Nasal Douche (END01): 1 spray per nostril 2-6 times per day or as often as required
  Interventions: Drug: Xylometazoline Nasal Spray; Device: Ectoin Nasal Douche

INTERVENTIONS:
Drug: Xylometazoline Nasal Spray — Application of Xylometazoline Nasal Spray in accordance with the instructions for use
  Other Names: NasenSpray-ratiopharm Erwachsene (adults)
Device: Ectoin Nasal Douche — Application of Ectoin Nasal Douche (END01) in accordance with the instructions for use
  Other Names: END01
  Groups: Xylometazoline + Ectoin Nasal Douche

SUMMARY:
The goal of this non interventional study is to investigate the efficacy, tolerability and safety of the newly developed Ectoin Nasal Douche END01. Within the study, END01 will be used as concomitant therapy in addition to the use of a Xylometazoline-containing decongestant nasal spray.

It will be investigated if the dosis of the used decongestant nasal spray might be reduced, the development of the disease might be positively influenced and/or the potentially occuring side effects (e.g. dryness of the nasal mucosa, sneezing) might be alleviated by using the Ectoin Nasal Douche as concomitant therapy.

DETAILED DESCRIPTION:
The current non-interventional study aims to investigate the efficacy, tolerability and safety of a decongestant Xylometazoline-containing nasal spray in comparison to use of a decongestant Xylometazoline-containing nasal spray together with an Ectoin-containing nasal douche in patients with acute viral rhinosinusitis.

Efficacy will be studied by documentation of the following symptoms:

* oedema, redness (assessed by rhinoscopy)
* nasal obstruction, nasal secretion, headache/face pain, loss of sense of smell/taste
* sore throat, cough

In parallel, participating patients will document their symptoms and the their quality of life over the entire study duration in patient diaries.

Patients of both genders aged 6 years and above can take part in the study if diagnosed with acute viral rhinosinusitis. The assignment of a patient to a particular treatment is not decided in advance but falls within current practice, and is clearly separated from the decision to include the patient into the study.

Study therapy will be applied in accordance with the respective instructions for use.

Study duration is 7-14 days, depending on the improvement of symptoms. At the end of the study, both the investigators and the patients are asked to judge the efficacy and tolerability of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute viral rhinosinusitis
* presence of common cold symptoms

Exclusion Criteria:

* contraindications in accordance with instructions for use
* acute bacterial rhinosinusitis
* chronic rhinosinusitis

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged above 6 years diagnosed with acute viral rhinosinusitis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Physicians' assessment of change of intensity of rhinosinusitis symptoms | day 0 and day 7 and (if necessary, depending on study duration) and on day 14
  Both on day 0 and on day 7 (and, if necessary, depending on study duration, on day 14), the physicians will assess rhinosinusitis symptoms oedema, redness of the nose, nasal obstruction, nasal secretion, facial pain/headache, smell/taste dysfunction and the concomitant symptoms dryness of the nasal mucosa and sore throat. Assessment will be carried out based on a 5-point scale (0=none to 4=very strong). Change of symptoms will be assessed comparing symptom scores on day 7 (or day 14, if applicable) to day 0. The investigators will use rhinoscopy, physical examination and interview of the patients for the assessments.

SECONDARY OUTCOMES:
Physicians' assessment of general well-being of patients | day 0 and day 7 and day 14 (if necessary, depending on study duration)
  The investigators will assess the well-being of patients using a 4-point scale (good condition to strong illness).
Patients' assessment of intensity of symptoms and their influence on quality of life | 7 to 14 days (depending on study duration)
  Patients will document their rhinosinusitis symptoms and their influence on quality of life (22 parameters in accordance with the "sino-nasal outcome test-22 questionnaire") and the additional symptom "dry nose". They will document their judgement daily in a patient diary using a 6-point scale (0=no problem to 5=as bad as possible).
Assessment of the efficacy of treatments | day 7 or day 14 (depending on study duration)
  At the end of the study, both investigators and patients will judge the overall efficacy of the treatment based on a 6-point scale (1=very good to 6=unsatisfactory).
Assessment of the tolerability of treatments | day 7 or day 14 (depending on study duration)
  Both investigators and patients will judge the tolerability of the treatments at the end of the study. Both investigators and patients will judge the tolerability based on a 6 point scale (1=very good to 6 = unsatisfactory).
Incidence of adverse events/serious adverse events | 7 to 14 days (depending on study duration)
  All occurring adverse events/serious adverse events will be documented during the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bilstein, Dr., Study Director — CSO
Locations (1):
- bitop AG, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided